CLINICAL TRIAL: NCT03673241
Title: A Randomized, Non-Blinded Clinical Trial of a Non-Invasive Perfusion Enhancement System (Guardian System) on Motor Recovery and Impact on Length of Stay in Mobility Impaired Ischemic Stroke Patients
Brief Title: Study of the Guardian System on Motor Recovery and Impact on Length of Stay in Ischemic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TurnCare Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-6235
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Motor Recovery; Length of Stay Reduction
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, non-blinded, randomized trial. This cohort will be divided into two groups: (1) The Control Group (2) The Study Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control Group (No Intervention): The Control Group will receive the standard support surface mattresses/bed surfaces and recovery chairs without the non-invasive perfusion enhancement system (The Guardian System)
- Study Arm (Experimental): The Study Arm will have the non-invasive perfusion enhancement system placed on their beds and recovery chairs. Patients will be utilizing the systems while lying in bed or sitting in the chair.
  Interventions: Device: Guardian System

INTERVENTIONS:
Device: Guardian System — The Study arm will have the Guardian system applied to their bed and recovery chair with the intent for the patient to have the inflatable surface utilized underneath them .
  Arms: Study Arm

SUMMARY:
This is a non-blinded randomized study that will investigate whether the use of a novel, non-invasive perfusion enhancement system (The Guardian System) impacts motor recovery and hospital length of stay in acute ischemic stroke patients.

DETAILED DESCRIPTION:
This clinical research study is a prospective, non-blinded randomized clinical trial. The study protocol and consent form have been approved by the IRB at the Study Institution. As per the study design, consecutive adult patients admitted to the neuro-intensive care unit, with acute ischemic stroke, meeting the inclusion and exclusion criteria will be consented and enrolled in the study. Both the Study and Control groups will receive the standard of care for ischemic stroke according to the hospitals' protocols, policies and procedures. After obtaining informed consent, patients in the study arm will have the non-invasive perfusion enhancement system (The Guardian System) placed on their beds and chairs. The inflatable surfaces (the enhancers) will be placed directly on the mattress and chair under the fitted sheet and bed linens. They will be secured with a non-porous, non-slip silicone attacher. An adaptive pressure controller will be attached to the perfusion enhancer through a connector set. The adaptive pressure controller will be secured to the bed foot board or side rail and have the ability to be secured to an Intravenous pole as necessary. Specific data points for each patient in the Experimental group will be entered into the Controller: they include the patient's weight in kilograms and the patient's position (bed or chair).

This study seeks to evaluate the device's effect on motor recovery and length of stay in a homogeneous ischemic stroke population that will be randomized for use of the novel non-invasive perfusion enhancement device from admission to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Only Acute Ischemic Stroke Patients
* Baseline Modified Rankin Score of less than or equal to 0-2
* Remains hemiplegic (left or right) with motor component score on National Institute of Stroke Health Scale of 2-4 on arm/leg with or without thrombectomy/tissue plasminogen activator
* Insured (Medicare or private)

Exclusion Criteria:

* Dementia or Alzheimer Diagnosis
* Concurrent hemodialysis
* Obesity with Body Mass Index greater than 33
* Baseline Modified Rankin Score of 3 to 5
* Patients requiring ventilator support of greater than 2 days
* Peripheral neuropathy
* Concurrent deep vein thrombosis or venous thromboembolism
* Presence of concurrent pre-existing pressure injury
* Prolonged inconsistent use of perfusion therapy defined as two or more consecutive hours off of the perfusion enhancement device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-03-28 (Estimated)

PRIMARY OUTCOMES:
Length of Stay Reduction in Acute Ischemic Stroke Patients in the Control and Study Arm Groups | The time frame will be up to and including 24 months
  The length of stay of acute ischemic stroke patients measured from the time of randomization until the the date of discharge or date of death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Fern Cudlip, MSN FNP CNRN, Principal Investigator — Good Samaritan Hospital
Locations (1):
- Good Samaritan Hospital, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakhan SE, Kirchgessner A, Hofer M. Inflammatory mechanisms in ischemic stroke: therapeutic approaches. J Transl Med. 2009 Nov 17;7:97. doi: 10.1186/1479-5876-7-97. PMID 19919699
- [Background] Bharucha JB, Seaman L, Powers M, Kelly E, Seaman R, Forcier L, McGinnis J, Nodiff I, Pawlak B, Snyder S, Nodiff S, Patel R, Squitieri R, Wang L. A Prospective Randomized Clinical Trial of a Novel, Noninvasive Perfusion Enhancement System for the Prevention of Hospital-Acquired Sacral Pressure Injuries. J Wound Ostomy Continence Nurs. 2018 Jul/Aug;45(4):310-318. doi: 10.1097/WON.0000000000000450. PMID 29889718
- [Background] Doll DN, Barr TL, Simpkins JW. Cytokines: their role in stroke and potential use as biomarkers and therapeutic targets. Aging Dis. 2014 Oct 1;5(5):294-306. doi: 10.14336/AD.2014.0500294. eCollection 2014 Oct. PMID 25276489
- [Background] Davies CA, Loddick SA, Toulmond S, Stroemer RP, Hunt J, Rothwell NJ. The progression and topographic distribution of interleukin-1beta expression after permanent middle cerebral artery occlusion in the rat. J Cereb Blood Flow Metab. 1999 Jan;19(1):87-98. doi: 10.1097/00004647-199901000-00010. PMID 9886359
- [Background] Zheng Z, Yenari MA. Post-ischemic inflammation: molecular mechanisms and therapeutic implications. Neurol Res. 2004 Dec;26(8):884-92. doi: 10.1179/016164104X2357. PMID 15727272
- [Background] Nour M, Scalzo F, Liebeskind DS. Ischemia-reperfusion injury in stroke. Interv Neurol. 2013 Sep;1(3-4):185-99. doi: 10.1159/000353125. PMID 25187778
- [Background] Du T, Zhu YJ. The regulation of inflammatory mediators in acute kidney injury via exogenous mesenchymal stem cells. Mediators Inflamm. 2014;2014:261697. doi: 10.1155/2014/261697. Epub 2014 Apr 15. PMID 24839354
- [Background] Jiang LP, Tu Q, Wang Y, Zhang E. Ischemia-reperfusion injury-induced histological changes affecting early stage pressure ulcer development in a rat model. Ostomy Wound Manage. 2011 Feb;57(2):55-60. PMID 21350273
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429